CLINICAL TRIAL: NCT03983031
Title: Rituximab - Immunotherapy for Obsessive-compulsive Disorder: An Open Pilot Study
Brief Title: Rituximab for Obsessive-compulsive Disorder. (RITS-PO-2019)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Region Örebro County (Other)
Collaborators: Örebro University, Sweden (Other)
Responsible Party: Principal Investigator, Susanne Bejerot, Principal investigator, Region Örebro County
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: EudraCT Number: 2018-004619-28
Record Dates: First submitted 2019-05-30; First posted 2019-06-12 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: Obsessive-Compulsive Disorder; Treatment Resistant Disorders
Keywords: Immunopsychiatry; pediatric acute-onset neuropsychiatric syndrome
MeSH Terms: conditions — Obsessive-Compulsive Disorder; Pediatric acute-onset neuropsychiatric syndrome | interventions — Rituximab

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Each patient will be video recorded at base line, week 12, 20 and 40 in order to enable blinded assessment by an independent rater, and for the patient's own evaluation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Rituximab — Infusion

SUMMARY:
This study evaluates the addition of rituximab to 12 patients diagnosed with treatment resistant obsessive-compulsive disorder in an open trial.

DETAILED DESCRIPTION:
Immunological factors may be determinants for some psychiatric disorders, thus immunomodulation may be helpful. Rituximab (antibodies against CD20, cluster of differentiation), a standard treatment for multiple sclerosis, is an anti-inflammatory drug, hitherto not tested for psychiatric disorders.

The aim of this study is to investigate whether the psychiatric symptoms of treatment-resistant adult psychiatric patients, diagnosed with obsessive-compulsive disorder (OCD), are significantly improved after treatment with rituximab. The investigator's purpose is to implement recent insights from "Immunopsychiatry" to find efficacious, but still tolerable treatment for these patients.

This is a single-site, 20-week, open pilot, add-on treatment as usual, trial, where the patients will be followed for 1 year.

Rituximab will be administered with one single dose of 1000 mg. Investigators will analyse inflammatory and metabolic biomarkers in relation to the primary outcome, treatment response (defined as clinically relevant reduction in the validated measure Y-BOCS). Other outcomes are "much" or "very much improved" on Clinical Global Impression - Improvement scale (CGI-I) and change in Personal and Social Performance Scale measuring overall disability.

ELIGIBILITY:
Inclusion Criteria (Swedish citizens):

1. patient ages 18 to 40 years.
2. a duration of illness exceeding 2 years.
3. correspond to "Markedly ill", "Severely ill" or "Among the most extremely ill patients" on the Clinical Global Impression - Severity scale (CGI-S).
4. Global Assessment of Functioning (GAF) below 50.
5. obsessive-compulsive disorder according to The Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5).
6. treatment resistance, i.e. failing to remit despite adequate treatments.
7. if female and with any risk for pregnancy, willing to use contraceptives.
8. if psychotropic treatment is prescribed the plasma concentrations of the drug must be tested and shown to be within therapeutic interval.
9. subjects should be judged by the investigator to be lucid and oriented to person, place, time, and situation when giving the informed consent.
10. immunoglobulin levels within the normal range.

Exclusion Criteria:

1. on-going immunomodulatory treatment.
2. pregnancy or breast-feeding.
3. weight below 40 kg.
4. clinically relevant on-going infection.
5. chronic infections .
6. positive screening test for hepatitis B, C, HIV or tuberculosis
7. any change of psychotropic medication within the previous 4 weeks
8. "much" or "very much" improved already at baseline according to CGI-I.
9. severe heart failure (NYHA grade IV) or other severe heart disease or history of cardiac arrhythmia or myocardial infarction.
10. unable to make an informed decision to consent to the trial.
11. in compulsory treatment.
12. treatment with clozapine within the last 2 months.
13. previous treatments with immunosuppressive agents.
14. malignancy currently or within 2 years prior to inclusion.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2019-08-08 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Yale-Brown obsessive- compulsive scale (Y-BOCS) | week 20
  Y-BOCS maps symptoms and measures severity of obsessive-compulsive symptoms by a clinician. Y-BOCS has a range between 0 and 40 points, higher scores denotes worse symptoms. Outcome is measured as change in Y-BOCS score from baseline. At least 35% reduction in the score since baseline is defined as a response.

SECONDARY OUTCOMES:
Personal and Social Performance Scale (PSP) | week 20
  Personal and Social Performance Scale (PSP) gives a score for disability. The PSP is a 100-point single-item rating scale (range 1-100), subdivided into 10 equal intervals. Lower scores denote lower functioning. The ratings are based mainly on the assessment of patient's functioning in four main areas: 1) socially useful activities; 2) personal and social relationships; 3) self-care; and 4) disturbing and aggressive behaviours. Change in score between enrolment and week 20 will be measured.
Clinical Global Impression-severity (CGI-S) scale | week 20
  CGI-S is a clinician rated measure of overall clinical severity that is rated on a scale between 1 and 7. A person with no clinical complaints or problems will get a score of 1. The score 7 indicates the highest level of severity is phrased as "Among the most extremely ill patients".
Clinical Global Impression-Improvement (CGI-I) in relation to inflammatory markers | week 20
  Clinical Global Impression-Improvement scale (CGI-I) measures change of symptoms on a 7 point Likert scale. A CGI-I score of 1 or 2 corresponds to be much or very much improved. Change in inflammatory markers in blood (gene expression and proteins) towards normality, in relation to clinical response (assessed by the clinician) will be measured.
Clinical Global Impression-Improvement (CGI-I). Proportion of responders. | week 20
  Clinical Global Impression-Improvement scale (CGI-I) measures change of symptoms on a 7 point Likert scale. A CGI-I score of 1 or 2 corresponds to be much or very much improved. Three different informants base their CGI-I evaluations on independent assessments: a) The treating clinician, b) The patient's self-assessment and c) A next of kin. If the mean value of these three is below 2.5 then the patient will be regarded as a responder (representing much or very much improved since baseline).
Clinical Global Impression-Improvement (CGI-I). | week 20
  Clinical Global Impression-Improvement scale (CGI-I) measures change of symptoms on a 7 point Likert scale. A CGI-I score of 1 or 2 corresponds to be much or very much improved. Three different informants base their CGI-I evaluations on independent assessments: a) The treating clinician, b) The patient's self-assessment and c) A next of kin. Range 3-21. A lower score depicts larger improvement.
Adverse event: Any Adverse Reactions (AAR). Safety and tolerability of Rituximab | week 20
  Any Adverse reactions (AAR) is a rating scale developed for this study and is not a validated questionnaire. It consists of a list of 26 symptoms. AAR maps adverse events related to rituximab treatment. These items are assessed for severity on a Likert scale (4 levels: none; mild; moderate; severe) and frequency (3 levels: occasionally; daily; several times daily). AAR is assessed by the clinician. An adverse event scale was required as an outcome measure by the Swedish Medical Products Agency.

OTHER OUTCOMES:
Yale-Brown obsessive- compulsive scale (Y-BOCS) | week 40
  Y-BOCS maps symptoms and measures severity of obsessive-compulsive symptoms by a clinician. Y-BOCS has a range between 0 and 40 points, higher scores denotes worse symptoms. Outcome is measured as change in Y-BOCS score from baseline. At least 35% reduction in the score since baseline is defined as a response.
Personal and Social Performance Scale (PSP) | week 40
  Personal and Social Performance Scale (PSP) gives a score for disability. The PSP is a 100-point single-item rating scale (range 1-100), subdivided into 10 equal intervals. Lower scores denote lower functioning. The ratings are based mainly on the assessment of patient's functioning in four main areas: 1) socially useful activities; 2) personal and social relationships; 3) self-care; and 4) disturbing and aggressive behaviours. Change in score between enrolment and week 40 will be measured.
Clinical Global Impression-severity (CGI-S) scale | week 40
  CGI-S is a clinician rated measure of overall clinical severity that is rated on a scale between 1 and 7. A person with no clinical complaints or problems will get a score of 1. The score 7 indicates the highest level of severity is phrased as "Among the most extremely ill patients".
Clinical Global Impression-Improvement (CGI-I) in relation to inflammatory markers | week 40
  Clinical Global Impression-Improvement scale (CGI-I) measures change of symptoms on a 7 point Likert scale. A CGI-I score of 1 or 2 corresponds to be much or very much improved. Change in inflammatory markers in blood (gene expression and proteins) towards normality, in relation to clinical response (assessed by the clinician) will be measured.
Changes in cognitive functioning | week 20
  Improvement in cognitive tests using a subset of tests included in Wechsler Adult Intelligence Scale (WAIS) (i.e. Block design, digit span, letter number sequencing and digit symbol coding, visuospatial test).
CGI-I in relation to treatment and evaluated by the treating clinician, the patient's self-assessment and a next of kin | week 40
  Clinical Global Impression-Improvement scale (CGI-I) measures change of symptoms on a 7 point Likert scale. A CGI-I score of 1 or 2 corresponds to be much or very much improved. Three different informants base their CGI-I evaluations on independent assessments: a) The treating clinician, b) The patient's self-assessment and c) A next of kin. Range 3-21. A lower score depicts larger improvement.
B cell subpopulations in relation to clinical response | week 20
  B-cell depletion at week 5, and B-cell subpopulations at week 20 in relation to clinical response (CGI-I) (assessed by the clinician) and baseline levels of B-cells.
Life quality measured with Brunnsviken Brief Quality of Life Scale (BBQ) | week 40
  BBQ is a 12-item self-rated measurement of life satisfaction, it is a likert scale, range 0-48. Higher scores denote higher life satisfaction.
Clinical Global Impression-Improvement (CGI-I). Proportion of responders. | week 40
  Clinical Global Impression-Improvement scale (CGI-I) measures change of symptoms on a 7 point Likert scale. A CGI-I score of 1 or 2 corresponds to be much or very much improved. Three different informants base their CGI-I evaluations on independent assessments: a) The treating clinician, b) The patient's self-assessment and c) A next of kin. If the mean value of these three is below 2.5 then the patient will be regarded as a responder (representing much or very much improved since baseline).

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Bejerot, MD, Principal Investigator — Region Örebro län
Locations (2):
- Sweden (2):
  - Region Örebro län, Örebro
  - Region Örebro Län, Örebro

IPD SHARING:
Plan to Share IPD: No
Details that can identify the patients will not be shared.